CLINICAL TRIAL: NCT03308006
Title: Knee Osteoarthritis Treatment With Adipose-derived Stem Cells: Phase II Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2018-04
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cells therapy (Experimental)
  Interventions: Biological: Stem cells

INTERVENTIONS:
Biological: Stem cells — Participants will be exposed to e abdominal liposuction procedure under local anesthesia for stem cells harvesting. Stem cells will be separated from fat cells in the adipose tissue then activated in Tissue Culture Lab at Research Center- Jeddah. The activated stem cells will be injected into the knee joint via 22G spinal needle. The intra-articular stem cells injections will be performed under Ultrasound guidance at the theater under spinal anesthesia. Each patient will receive 1.0× 108 stem cells in 3 mL of normal saline.

SUMMARY:
In 1990, the prevalence of osteoarthritis of the hip or knee was very low 3.5% in Saudi Arabia, it increased to 53.3% and 60.9% in male in female patients respectively in 2002. The existing management of OA is conservative and pharmacological management aiming to relief symptoms of osteoarthritis and improves joint function. Results of a Meta-Analysis showed that mesenchymal stem cell is effectiveness and safe to treat knee osteoarthritis. In 1990, the prevalence of osteoarthritis of the hip or knee was very low 3.5% in the Kingdom of Saudi Arabia and it increased to 53.3% and 60.9% in male in female patients respectively in 2002. Results of a Meta-Analysis showed that mesenchymal stem cell is effectiveness and safe to treat knee osteoarthritis. This study will be a single center phase II-one arm clinical trial. It will be conducted at KF SH&RC-Jeddah. 18 participants will be recruited from orthopedic clinics. Participate will be evaluated before inclusion in the study. Participants will be exposed to e abdominal liposuction procedure under local anesthesia for stem cells harvesting. Stem cells will be separated from fat cells in the adipose tissue then activated in Tissue Culture Lab at Research Center- Jeddah. The activated stem cells will be injected into the knee joint via 22G spinal needle. The intra-articular stem cells injections will be performed under Ultrasound guidance at the theater under spinal anesthesia. Each patient will receive 1.0× 108 stem cells in 3 mL of normal saline

DETAILED DESCRIPTION:
STUDY DESIGN, LOCATION AND PATIENTS This study will be a single center phase II one arm clinical trial. It will be conducted at King Faisal Specialist Hospital &Research Center (Gen. Org.)-Jeddah. The decided sample size will be between 12 to 18 participants. Participants will be recruited from orthopedic clinics. Each patient will receive 1.0× 108 stem cells in 3 mL of normal saline.

All patients who are potentially eligible to be included in the study, and agreed to participate will be evaluated medically. Baseline assessment will involve complete general and orthopedic physical examination. Complete laboratory investigations and radiological investigations including diagnostic MRI of the knee to confirm the diagnosis will performed to each patient.

Inclusion Criteria In this study, participants will be considered as having Knee osteoarthritis if the patient's x-rays showed grade 2 or higher Kellgren and Lawrence scale. He/she will be potentially eligible to be included in the study if his/her age is between 45 and 65 years and diagnosed by orthopedic consultant as having idiopathic osteoarthritis of the knee and had an average pain intensity of grade 4 or more on a 10-point visual analog for at least one year.

Exclusion Criteria Patient will be excluded if she/he had history of chronic rheumatic or inflammatory diseases, poorly controlled diabetes, or currently on OA treatments.

Data collection Potentially eligible participants will receive verbal and formal written information about the study and invited to participate. Eligible participants who provide written consent to participate will be asked to fill out a well known reliable and valid Musculoskeletal Pain Questionnaire (The Orebro Musculoskeletal Pain Questionnaire).

Procedures The procedure of KOA stem cell therapy will be done in four stages, harvesting, separation, activation, and treatment stage. In summary, Participants in this phase II one arm clinical trial will be exposed to simple abdominal liposuction procedure under local anesthesia for stem cells harvesting. Stem cells will be separated from fat cells in the adipose tissue then activated in Tissue Culture Lab at Research Center- JEDDAH after that the activated stem cells will be injected into the knee joint via 22G spinal needle. The intra-articular stem cells injections will be performed under Ultrasound guidance at the theater under spinal anesthesia.

Personnel Simple abdominal Liposuction will be performed by accredited plastic surgeon. Qualified scientist and qualified and trained technicians will perform stem cells separation and activation under good manufacturing practice conditions, and orthopedic surgeon will perform intra-articular stem cells injections.

Outcome Measures Participants will be followed for one year after the date of stem cells knee joint injection and monitored and evaluated for serious adverse events, clinical outcomes, the size, depth and histological assessment of regenerated cartilage.

Statistical Analysis Categorical data will be summarized by measuring the frequency and percentage and measures of central tendency and dispersions will be used summarize numeric data. Paired t test and Wilcoxon signed rank test will be used to compare the changes from baseline in parametric and non-parametric data respectively. The analysis will be performed using SPSS version 16

ELIGIBILITY:
Inclusion Criteria:

* age between 45 and 65.
* Participants having Knee osteoarthritis grade 2 or higher "Kellgren and Lawrence scale"
* Participants had an average pain intensity of grade 4 or more on a 10-point visual analog for at least one year.

Exclusion Criteria:

* Patient with history of rheumatic or chronic inflammatory diseases
* Patient poorly controlled diabetes,
* Patient who currently on OA treatment such as corticosteroids, chondroitin sulfate, glucosamine or hyaluronic acid.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Regenerated cartilage | One year
  Histological assessment of regenerated cartilage

CONTACTS AND LOCATIONS:
Overall Officials: . Zainullah Al Shareef, MD, Study Chair — King Faisal Specialist Hospital & Research Cener -Jeddah
Locations (1):
- King Faisal Sepcialist Hospital and Research Center, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No